CLINICAL TRIAL: NCT01005173
Title: Identification of New Mechanistic Biomarkers of Adverse Response to Acetaminophen
Brief Title: Acetaminophen Biomarkers
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1R01DK081406-01A1 (NIH); 1 R01 DK081406-01A1 - NIH
Record Dates: First submitted 2009-10-28; First posted 2009-10-30 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Acetaminophen Toxicity
Keywords: Acetaminophen; APAP

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group A: Subjects receiving recommended doses of acetaminophen in the hospital. 140 Subjects
- Group B: Healthy Volunteers - No acetaminophen exposure within 14 days of enrollment 23 Subjects
- Group C: Acetaminophen Overdose Subjects - Hospitalized 90 Subjects

SUMMARY:
This study is a non-intervention, multicenter study to address biomarkers of acetaminophen toxicity in children. Specifically, the study will examine acetaminophen (APAP) protein adducts and markers of liver injury in the blood samples of hospitalized children and adolescents who are receiving standard doses of acetaminophen, and children and adolescents who are status post acetaminophen overdose. Ultimately, the data generated from this study will be used to establish second generation biomarkers of acetaminophen toxicity, based on specific adduct proteins, which can be used in future risk assessment studies of children receiving acetaminophen.

ELIGIBILITY:
Inclusion Criteria:

Group A:

* Children ages 1-18 inclusive
* Hospitalized children who are likely to receive or are receiving recommended doses of APAP

Group B:

* Children ages 1-18 inclusive
* Children with no APAP use in the past 14 days

Group C:

* Children ages 1-18 inclusive
* Hospitalized from an acute overdose of APAP
* Time of APAP overdose is known or can be estimated within a two hour window

Exclusion Criteria:

Group A:

* Acute or chronic APAP overdose within 14 days
* Known history of liver disease or dysfunction

Group B:

* APAP within the last 14 days
* Known history of liver disease or dysfunction

Group C:

* Chronic overdoses of APAP, defined as multiple time point ingestions of APAP
* History of previous APAP overdose
* Known pre-existing liver disease

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children Ages 1-18
  Group A - Hospitalized receiving acetaminophen
  Group B - Healthy volunteers - no acetaminophen within 14 days
  Group C - Acetaminophen Overdose - Hospitalized
Sampling Method: Non-Probability Sample
Enrollment: 253 (Estimated)
Dates: Start 2009-08; Primary Completion 2018-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Laura P James, MD, Principal Investigator — Arkansas Children's Hospital Research Institute
Locations (8):
- United States (8):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Kosair Charities Pediatric Clinical Research Unit University of Louisville, Louisville, Kentucky
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Akron Children's Research Center, Akron, Ohio
  - University of Toledo Health Science Center, Toledo, Ohio
  - Cook's Children's Health System, Fort Worth, Texas
  - Baylor College of Medicine - Texas Children's Hospital, Houston, Texas